CLINICAL TRIAL: NCT02923869
Title: Comparative Study Between Levobupivacaine and Bupivacaine for Nerve Block During Pediatric Primary Cleft Palate Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MOHAMED F. MOSTAFA, Lecturer of Anesthesia and Intensive Care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SMB Levobupivacaine
Record Dates: First submitted 2016-09-30; First posted 2016-10-05 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Recovery After Cleft Palate Surgery
Keywords: Levobupivacaine; Bupivacaine; Nerve Block; Cleft Palate
MeSH Terms: conditions — Cleft Palate | interventions — Levobupivacaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group L (Active Comparator): Children will receive 0.15 ml/kg of 0.2% Levobupivacaine
  Interventions: Drug: Levobupivacaine
- Group B (Active Comparator): Children will receive 0.15 ml/kg of 0.2% Bupivacaine
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Levobupivacaine — Children will receive 0.15 ml/kg of 0.2% Levobupivacaine through bilateral suprazygomatic MNB.
  Arms: Group L
Drug: Bupivacaine — Children will receive 0.15 ml/kg of 0.2% Bupivacaine through bilateral suprazygomatic MNB.
  Arms: Group B

SUMMARY:
A cleft deformity of the lip and/or palate is one of the commonest major birth defects.

Primary surgery of cleft palates (CP) varies according to the different surgical teams. Its peculiarity lies in the numerous care management protocols proposed according to the surgical techniques used, operating time (between M3 and M18 of life), anesthetic technique and postoperative management.

This surgery must be associated to a specific care management because of potential associated complications, especially the risk of obstruction of the upper respiratory tract and respiratory distress majored by the use of morphine anesthetics during and after surgery.

Adequate postoperative analgesia in children is a vital part of perioperative care. Regional block given preoperatively in combination with general anesthesia (GA) provides good preemptive analgesia. It is associated with perioperative hemodynamic stability, rapid and complete recovery and reduced analgesic requirement in the postoperative period.

CP repair is painful, necessitating high doses of intravenous (IV) opioids. Therefore, the risk of postoperative respiratory depression and airway obstruction is important, and continuous monitoring is required during the initial 24-h postoperative period. Cleft palate surgery is not only painful, but may also compromise the airway, particularly in children with craniofacial syndromes. Opiate analgesia has the potential to further compromise the airway, whereas bilateral maxillary nerve block can provide analgesia without the risk of respiratory depression in these vulnerable patients. Bilateral maxillary nerve block is performed using a suprazygomatic approach and is based on a computer tomography study.

The nerve supply to the hard and soft palate is from the greater and lesser palatine nerves passing through the sphenopalatine ganglion. The maxillary nerve (MN) provides sensory innervation of the anterior and posterior palate, the upper dental arch, the maxillary sinus, and the posterior nasal cavity. Maxillary nerve block (MNB) through the infrazygomatic route, used for the treatment of trigeminal neuralgia in adults, permits anesthesia of the entire palatine territory. However, this nerve block has led to complications such as orbital puncture, intracranial injection, maxillary artery puncture, or posterior pharyngeal wall injury.

DETAILED DESCRIPTION:
A prospective randomized controlled double blind study using a computer generated randomization scheme will be conducted in Assiut University Hospitals and will be carried out on 60 children undergoing primary cleft palate repair surgery. Combined general anesthesia and regional bilateral maxillary nerve block (MNB) will be used for anesthesia in these surgeries.

The study drugs (used in MNB) and randomization will be prepared by the second anesthetist. The MNB and observed parameters (intraoperative and postoperative) will be done by the first anesthetist.

Children will be randomly allocated into one of two groups of 30 patients each:

Group L: children will receive 0.15 ml/kg of 0.2% Levobupivacaine

Group B: children will receive 0.15 ml/kg of 0.2% Bupivacaine

Preoperative Assessment

The day prior to surgery, all children participating in this study will undergo pre-anesthetic checkup (preoperative fitness) including detailed history from the parents, thorough general, physical and systematic examinations. Weight and height of all children will be carefully recorded.

Anesthetic Technique

Premedication: All children will be premedicated with intramuscular midazolam 0.05 mg/kg 10-20 minutes before induction of general anesthesia.

Monitoring: Pulse Oxymetry (SaO2), Non-Invasive Mean Arterial Blood Pressure (MABP), ECG, End Tidal CO2 (EtCO2) and Non-Invasive Temperature probes will be applied to each patient.

After 3 minutes of 100% pre-oxygenation, general anesthesia will be induced by Sevoflurane inhalation 4-6% MAC via facemask then intravenous line will be secured and intravenous fluids (NaCl 0.9%) will be started at the calculated volume and rate. Fentanyl 1 µg/kg and Propofol 1.5 mg/kg will be given intravenously then intubation with oral RAE tube of the appropriate size will be inserted and secured. Assisted ventilation will be adjusted to maintain 30-35 mmHg EtCO2. Anesthesia will be maintained with 100% O2 and Sevoflurane 2-4% MAC. Broad spectrum antibiotic will be given to each child participated in the study.

Suprazygomatic MNB: Bilateral suprazygomatic MNB will be performed after complete aseptic preparation of the skin and before surgery in an anesthetized patient. Success of MNB will be assessed by the lack of sympathetic response to surgical stimulation.

Data Collection

Demographic data: including age, sex, weight and height.

Intraoperative data: heart rate (HR), mean arterial pressure (MAP), ECG, SaO2, EtCO2 and Sevoflurane MAC % will be measured every 15 minutes after MNB till the end of the surgery.

Postoperative data: HR, MAP, SaO2 and respiratory rate (RR) will be measured at the same times of pain assessment times.

Pain Severity: pain will be assessed by the second anesthetist blinded to the study drug used. Pain score will be evaluated on arrival to recovery room (T0), 1, 2, 4, 6, 8, 12 and 24 hours using the FLACC pain scale (Face, Legs, Activity, Cry and Consolability scale). If FLACC score ≥ 3, IV nalbuphine 0.1 mg/kg will be given for supplemental analgesia.

Time of the first analgesic requirement, total dose of nalbuphine consumption or any adverse effects (sedation, vomiting, respiratory depression, bleeding at the puncture site or any systemic toxicity related to the local anesthetic) will also be recorded.

Sedation score: will be evaluated by the 4 points (1-4) score. (Awake and alert -1, Sedated and responding to verbal command-2, Sedated and responding to mild stimulus-3, Sedated and responding to moderate to severe physical stimulus-4).

Blood glucose level will be measured before MNB, 15 minutes after block and 2 hours after end of surgery.

Statistical Analysis

All data will be collected and processed using SPSS (SPSS Inc., Chicago, Illinois, USA) version 20. All results will be expressed as mean ± SD, range, numbers and percentages. Categorical data will be compared using Chi-Square test. Non parametric data will be compared using the Mann-Whitney U test. Numerical data will be compared using the Independent Samples Student t-Test. P ˂ 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-10 years
* Both sexes
* ASA I or II
* Primary cleft palate

Exclusion Criteria:

* Any allergy to local anesthetics
* Coagulation disorders
* Local infection or injury at site of MNB
* Concomitant rhinoplasty
* Associated other congenital anomalies
* History of upper or lower airway diseases
* History of sleep apnea

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
recovery after surgery | 2 hours
  sedation of the child in the recovery room will be monitored

SECONDARY OUTCOMES:
FLACC score | 24 hours
  Nalbuphine will be given when visual analogue score ≥ 3
Intraoperative and Postoperative Complications | 24 hours
  percentage of patients with any complications will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: HAMDY A YOUSSEF, MD, Study Chair — Assiut University
Locations (1):
- Assiut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided